CLINICAL TRIAL: NCT00622453
Title: A Registry of Arrhythmias in Myotonic Muscular Dystrophy
Brief Title: Arrhythmias in Myotonic Muscular Dystrophy
Acronym: DM1
Status: Completed | Type: Observational
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Muscular Dystrophy Association (Other)
Responsible Party: William Groh, MD, Indiana University
Organization: Indiana University (Other)
Other Study IDs: 9609-31
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Muscular Dystrophy; Arrhythmia; Sudden Cardiac Death
MeSH Terms: conditions — Muscular Dystrophies; Arrhythmias, Cardiac; Death, Sudden, Cardiac | interventions — Mass Screening; Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Registry of Arrhythmias: Screening of individuals with myotonic muscular dystrophy to evaluate the utility of non-invasive electrocardiographic screening methods and history in predicting serious arrhythmic events.
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — Electrocardiography Blood Test
  Other Names: ECG; Holter Monitor; Blood Test

SUMMARY:
Adult myotonic muscular dystrophy (Steinert's disease) is the most common inherited neuromuscular disorder. Cardiac rhythm disturbances occur frequently in this disease state and may be responsible for up to one-third of deaths. In this study, we intend to evaluate the utility of non-invasive electrocardiographic screening methods and history in predicting serious arrhythmic events.

DETAILED DESCRIPTION:
The long term objectives of this population study is a more defined natural history, optimal diagnostic testing methodology, and methods of therapy for arrhythmias in individuals with myotonic muscular dystrophy. The goal is a more adequate definition of appropriate diagnosis and therapy for arrhythmias in order to decrease the likelihood of cardiac morbidity and mortality in this disorder.

The specific aims of the study involve an initial survey of individuals with myotonic muscular dystrophy detailing multiple factors. Non-invasive electrocardiographic testing will be done. Using this initial data and subsequent follow-up data collected yearly the cohort of patients will be followed as to arrhythmia development over a minimum of five years and likely longer with a long-term registry and evaluation of National Death Records and Ancestry.com. This project is unique in that it characterizes a non-neurologic abnormality associated with a neuromuscular disease, myotonic muscular dystrophy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and over
2. Willing to sign informed consent
3. Have a previous diagnosis of myotonic muscular dystrophy

Exclusion Criteria:

1. Under age 18.
2. Unwilling to sign consent.
3. Unwilling to commit to long-term follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient Recruitment: Will take place at the 230 hospital-affiliated MDA neuromuscular clinics. Individuals with myotonic dystrophy will be identified in the MDA clinics these will be asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 448 (Actual)
Dates: Start 1996-09; Primary Completion 2006-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Evaluate incidence of arrhythmias in myotonic muscular dystrophy | 3 years

SECONDARY OUTCOMES:
Evaluate with diagnostic non-invasive electrocardiogram (ECG) | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: William Groh, MD, Principal Investigator — Indiana School of Medicine
Locations (1):
- Krannert Institute of Cardiology, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Groh WJ, Groh MR, Saha C, Kincaid JC, Simmons Z, Ciafaloni E, Pourmand R, Otten RF, Bhakta D, Nair GV, Marashdeh MM, Zipes DP, Pascuzzi RM. Electrocardiographic abnormalities and sudden death in myotonic dystrophy type 1. N Engl J Med. 2008 Jun 19;358(25):2688-97. doi: 10.1056/NEJMoa062800. PMID 18565861
- [Result] Bhakta D, Lowe MR, Groh WJ. Prevalence of structural cardiac abnormalities in patients with myotonic dystrophy type I. Am Heart J. 2004 Feb;147(2):224-7. doi: 10.1016/j.ahj.2003.08.008. PMID 14760317
- [Result] Hardin BA, Lowe MR, Bhakta D, Groh WJ. Heart rate variability declines with increasing age and CTG repeat length in patients with myotonic dystrophy type 1. Ann Noninvasive Electrocardiol. 2003 Jul;8(3):227-32. doi: 10.1046/j.1542-474x.2003.08310.x. PMID 14510658
- [Result] Groh WJ, Lowe MR, Zipes DP. Severity of cardiac conduction involvement and arrhythmias in myotonic dystrophy type 1 correlates with age and CTG repeat length. J Cardiovasc Electrophysiol. 2002 May;13(5):444-8. doi: 10.1046/j.1540-8167.2002.00444.x. PMID 12030525
- [Derived] Bhakta D, Shen C, Kron J, Epstein AE, Pascuzzi RM, Groh WJ. Pacemaker and implantable cardioverter-defibrillator use in a US myotonic dystrophy type 1 population. J Cardiovasc Electrophysiol. 2011 Dec;22(12):1369-75. doi: 10.1111/j.1540-8167.2011.02200.x. Epub 2011 Oct 28. PMID 22035077
- [Derived] Bhakta D, Groh MR, Shen C, Pascuzzi RM, Groh WJ. Increased mortality with left ventricular systolic dysfunction and heart failure in adults with myotonic dystrophy type 1. Am Heart J. 2010 Dec;160(6):1137-41, 1141.e1. doi: 10.1016/j.ahj.2010.07.032. PMID 21146669